CLINICAL TRIAL: NCT00513071
Title: A Phase II Trial of AZD0530 in Hormone Refractory Prostate Cancer (HRPC)
Brief Title: AZD0530 in Treating Patients With Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02842; PHII-79; N01CM62209 (NIH); N01CM62201 (NIH); CDR0000559142 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-03

CONDITIONS: Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — saracatinib

ARMS (1):
- Treatment (saracatinib) (Experimental): Patients receive oral AZD0530 once daily. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: saracatinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: saracatinib — Given orally
  Other Names: AZD0530
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well AZD0530 works in treating patients with prostate cancer that did not respond to hormone therapy. AZD0530 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypothesis that AZD0530 will improve the prostate-specific antigen (PSA) response rate and progression-free survival (PFS) in comparison with historical controls for patients with hormone-refractory prostate cancer (HRPC).

II. Evaluate the time to treatment failure and overall survival of patients with HRPC treated with AZD0530.

III. Evaluate the toxicities and tolerance of AZD0530 therapy in the HRPC population.

OUTLINE: This is a multicenter study.

Patients receive oral AZD0530 once daily. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for the first 2 years and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer with a Gleason score available or interpretable and meeting 1 of the following criteria:

  * No prior chemotherapy and relatively minimal cancer spread
  * Only one prior taxane-based chemotherapy for aggressive and/or symptomatic disease
* Must have prostate cancer considered to be hormone refractory or androgen independent by one or more of the following criteria (despite androgen deprivation and anti-androgen withdrawal when applicable):

  * Progression of unidimensionally measurable disease assessed within 28 days prior to initial administration of drug
  * Progression of evaluable but not measurable disease assessed within 28 days prior to initial administration of drug for PSA evaluation and within 42 days for imaging studies (e.g., bone scans)
* Patients must have nonmeasurable disease (e.g., nuclear medicine bone scans) and non-target lesions (e.g., PSA level) assessed within 28 days prior to initial administration of drug

  * Measurable disease is not required but is allowed
* Must be surgically or medically castrated

  * If the method of castration was luteinizing hormone-releasing hormone (LHRH) agonists (e.g., leuprolide or goserelin), then the patient must be willing to continue the use of LHRH agonists
  * Serum testosterone must be at castrate levels (< 50 ng/dL) at least 3 months prior to registration
* ECOG performance status 0-2
* WBC >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin > 9 g/d
* Total bilirubin within normal institutional limits
* AST/ALT =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min
* Must agree to use adequate contraception prior to study entry and for the duration of study participation
* At least 3 weeks since the completion of chemotherapy and radiotherapy and the patient must have recovered from the side effects of the therapy
* At least 28 days since prior non-steroidal anti-androgens (e.g., flutamide) (42 days for bicalutamide or nilutamide) or hormonal treatment (e.g., ketoconazole) and demonstrated progression of disease since the agents were suspended
* Concurrent bisphosphonate therapy is allowed

Exclusion Criteria:

* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biological composition to AZD0530
* Patients with any of the following conditions that impair the ability to swallow AZD0530 tablets

  * Gastrointestinal tract disease resulting in an inability to take oral medication or requiring IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Use of specifically prohibited CYP3A4-active agents or substances

  * Prohibited drugs should be discontinued 7 days prior to the administration of the first dose of AZD0530 and for 7 days following discontinuation of AZD0530
* Patients receiving any other investigational agents
* No investigational or commercial agents or therapies other than study drugs may be administered with the intent to treat the patient's malignancy
* HIV-positive patients on combination antiretroviral therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo Lara, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Saracatinib): Patients receive oral AZD0530 at 175 mg once daily. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  saracatinib: Given orally
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Saracatinib)
Started | 28
Completed | 23
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 67 [50 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate
Description: Complete Response (CR), disappearance of all measurable and non-measurable disease. No new lesions. PSA ≤ 0.2 ng/mL; Partial Response (PR), a decline in PSA by at least 30%, confirmed by a second PSA value four or more weeks later; Overall Response (OR) = CR + PR
Time Frame: PSA measured every 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 28
percentage of participants | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS defined as time between start of treatment and disease progression or death. Using the method of Kaplan-Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From start of treatment until progression or death, up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 28
Months | 1.9 [1.8 to 3.7]

3. Secondary Outcome: Time to Treatment Failure
Description: Defined as the time from start of treatment to the discontinuation of treatment for any reason, including disease progression, treatment toxicity, patient preference, or death Will be summarized using the Kaplan-Meier product-limit estimators. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From first day of treatment until discontinuation of treatment, up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 28
Months | 1.9 [1.7 to 2.2]

4. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: From start of treatment, up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 28
Months | 26.0 [19.8 to 61.7]

5. Secondary Outcome: Toxicity Data
Description: Toxicity assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. All grade 3 or worse toxicities (Possibly, Probably, or Definitely) attributed to AZD0530.
Time Frame: Up to 2 years
Population: One patient died unexpectedly at home. No autopsy was performed. Treatment was listed as possible cause along with diabetes mellitus, morbid obesity, hypertension, hypercholesterolemia, and renal failure.
Measure: Number; unit: participants
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 28
participants
  Grade 3 : Alanine aminotransferase (ALT) | 1
  Grade 3 : Asparate aminotransferase (AST) | 1
  Grade 3 : Nausea | 1
  Grade 3 : Vomiting | 1
  Grade 3 : Lymphopenia | 1
  Grade 3 : Death, not associated with CTC term | 0
  Grade 5 : Alanine aminotransferase (ALT) | 0
  Grade 5 : Asparate aminotransferase (AST) | 0
  Grade 5 : Nausea | 0
  Grade 5 : Vomiting | 0
  Grade 5 : Lymphopenia | 0
  Grade 5 : Death, not associated with CTC term | 1

6. Secondary Outcome: Relationship Between Changes in Laboratory Correlates and Response and Survival
Time Frame: Up to 2 years
Population: Laboratory correlates were not collected.
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 0

7. Secondary Outcome: N-telopeptide and Deoxypyridinoline as Prognostic Bone Markers
Time Frame: At baseline, at 6 hours, at each course (day 1), and at 2 years
Population: Bone marker data was not collected.
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events over a 23 month time period.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Saracatinib)
All-Cause Mortality (participants affected / at risk) | 1/28
Serious Adverse Events (participants affected / at risk) | 5/28
Other Adverse Events (participants affected / at risk) | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Saracatinib) (N=28)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Saracatinib) (N=28)
Hemoglobin decreased (Blood and lymphatic system disorders) | 20 (33)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (9)
Diarrhea (Gastrointestinal disorders) | 7 (9)
Dyspepsia (Gastrointestinal disorders) | 2 (4)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5)
Chills (General disorders) | 3 (3)
Disease progression (General disorders) | 4 (4)
Edema limbs (General disorders) | 4 (4)
Fatigue (General disorders) | 13 (23)
Fever (General disorders) | 4 (5)
Flu-like symptoms (General disorders) | 1 (1)
General symptom (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (10)
Alkaline phosphatase increased (Investigations) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 16 (39)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 5 (8)
INR increased (Investigations) | 2 (3)
Leukocyte count decreased (Investigations) | 4 (6)
Lymphocyte count decreased (Investigations) | 6 (6)
Neutrophil count decreased (Investigations) | 2 (5)
Platelet count decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (2)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (9)
Blood glucose increased (Metabolism and nutrition disorders) | 10 (18)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 1 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 3 (3)
Serum calcium decreased (Metabolism and nutrition disorders) | 5 (5)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (2)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Abducens nerve disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 4 (5)
Urinary incontinence (Renal and urinary disorders) | 2 (3)
Urinary retention (Renal and urinary disorders) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less